CLINICAL TRIAL: NCT07122115
Title: The Effect of Mindfulness-Based Childbirth and Parenting Education on Birth Parameters and Postpartum Adaptation in Pregnant Women With Distress
Brief Title: Mindfulness-Based Childbirth Education for Pregnant Women With Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, MERVE GÜL TİREN, Specialist Nurse, PhD Candidate, Principal Investigator, Kayseri Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KayseriTRH-distress
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: PRENATAL DISTRESS
Keywords: MİNDFULNESS; PRENATAL DİSTRESS; FEAR OF CHILDBİRTH; MATERNAL ATTACHMENT

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups: an intervention group receiving mindfulness-based childbirth and parenting education, and a control group receiving standard prenatal care. Each group was followed independently throughout the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Prenatal Care (No Intervention): Participants in this group received routine prenatal care and standard childbirth education provided by the hospital without any mindfulness component.
- Experimental Arm (Experimental): Participants in this group received an 8-week mindfulness-based childbirth and parenting education program, including guided mindfulness practices, psychoeducation, and home assignments.
  Interventions: Behavioral: Mindfulness-Based Childbirth and Parenting Education

INTERVENTIONS:
Behavioral: Mindfulness-Based Childbirth and Parenting Education — The intervention was an 8-week mindfulness-based childbirth and parenting education program specifically adapted for pregnant women experiencing prenatal distress. The program included weekly 120-minute online sessions combining formal mindfulness practices (such as mindful breathing, body scan, and sitting meditation), informal exercises (e.g., mindful eating, mindful walking), psychoeducation, group sharing, and guided reflections.
  Participants were also asked to complete daily home practice assignments using audio recordings. The content was adapted from the Mindfulness-Based Childbirth and Parenting (MBCP) curriculum and integrated with prenatal education. The intervention was delivered by a trained instructor and tailored to meet the emotional and cognitive needs of expectant mothers.
  Arms: Experimental Arm

SUMMARY:
This randomized controlled trial aimed to evaluate the effects of a mindfulness-based childbirth and parenting education program on pregnant women experiencing prenatal distress. A total of 31 participants were randomly assigned to either an intervention group, which received an 8-week mindfulness-based education, or a control group, which received standard prenatal care. The study assessed outcomes such as pregnancy-related stress, fear of childbirth, conscious awareness, maternal attachment, and postpartum adaptation.

DETAILED DESCRIPTION:
This study was conducted to investigate the effects of a mindfulness-based childbirth and parenting education program on pregnant women who were identified as having prenatal distress. A randomized controlled trial design was used with a pre-test/post-test model. The participants were recruited from Kayseri City Training and Research Hospital's Pregnancy School and Outpatient Clinic between November and December 2022.

A total of 201 pregnant women were screened using the Tilburg Pregnancy Distress Scale (TPDS), and 31 women who scored 28 or higher and met the inclusion criteria were selected. Participants were randomly assigned into two groups: an intervention group (n=16) that received an 8-week mindfulness-based childbirth and parenting education program, and a control group (n=15) that received standard prenatal education.

The mindfulness-based program was conducted online and included guided mindfulness practices, psychoeducation, breathing exercises, and home assignments. Each session lasted approximately 120 minutes and was held once a week for eight consecutive weeks. Participants were also encouraged to practice formal and informal mindfulness exercises at home throughout the program.

The data were collected using several validated instruments, including the Tilburg Pregnancy Distress Scale, Mindful Attention Awareness Scale (MAAS), Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ), Visual Analog Scale (VAS) for labor pain, Maternal Attachment Scale, and Postpartum Self-Evaluation Questionnaire. Data collection occurred at multiple time points: before the intervention, after the intervention, on the first postpartum day, and during the first and fourth postpartum months.

ELIGIBILITY:
Inclusion Criteria:Female participants aged 18 to 35

First-time pregnancy (primigravida)

Gestational age between 24 and 32 weeks

No chronic medical or psychiatric conditions

Able to participate in online sessions

TPDS (Tilburg Pregnancy Distress Scale) score of 28 or higher

Minimum literacy level to understand consent and questionnaires

Voluntary participation and signed informed consent

-

Exclusion Criteria:

* High-risk pregnancy (e.g., preeclampsia, placenta previa)

Multiple pregnancy (e.g., twins or more)

Existing diagnosis of major psychiatric disorders

Participation in any previous mindfulness training

Inability to complete follow-up assessments

Non-consent or withdrawal from the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Prenatal Distress Level | From baseline (pre-intervention) to immediately post-intervention (approximately 8 weeks)
  Measured using the Tilburg Pregnancy Distress Scale (TPDS), which assesses pregnancy-related emotional distress.

SECONDARY OUTCOMES:
Change in Mindful Awareness | Baseline and post-intervention (8 weeks)
  Measured using the Mindful Attention Awareness Scale (MAAS). Higher scores indicate greater mindfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Training and Research Hospital, Kayseri, Kocasi̇nan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical concerns regarding participant privacy, as well as institutional restrictions on data sharing without explicit participant consent.

DOCUMENTS (1):
  • Study Protocol (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT07122115/Prot_000.pdf